CLINICAL TRIAL: NCT00709475
Title: Observational Safety Study in Subjects Using Levemir® (Insulin Detemir) for the Treatment of Type 2 Diabetes Mellitus
Acronym: LevSafeQD
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: NN304-3551
Record Dates: First submitted 2008-06-30; First posted 2008-07-03 (Estimated); Last update posted 2016-10-28 (Estimated); Status verified 2016-10

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — Insulin Detemir

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- A
  Interventions: Drug: insulin detemir

INTERVENTIONS:
Drug: insulin detemir — Start dose and frequency to be prescribed by the physician as a result of the normal clinical evaluation
  Other Names: Levemir®, NN304

SUMMARY:
This study is conducted in Asia. The aim of this observational study is to evaluate the incidence of serious adverse drug reactions while using insulin detemir under normal clinical practice conditions in the Gulf countries

ELIGIBILITY:
Inclusion Criteria:

* After the physician decision has been made to use insulin detemir therapy, any subject with Type 2 diabetes is eligible for the study, including newly-diagnosed subjects who have never received insulin or an insulin analogue before. The selection of the subjects will be at the discretion of the individual physician

Exclusion Criteria:

* Subjects who are unlikely to comply with protocol, e.g. uncooperative attitude, inability to return for the final visit;
* Subjects currently being treated with insulin detemir;
* Subjects who previously enrolled in this study or studies related to NovoMix 30;
* Subjects with a hypersensitivity to insulin detemir or to any of the excipients;
* Women who are pregnant, breast feeding or have the intention of becoming pregnant within next 8 months.

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Type 2 diabetic patients
Sampling Method: Probability Sample
Enrollment: 747 (Actual)
Dates: Start 2008-05; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Incidence of serious adverse drug reactions, evaluated via number of major hypoglycaemic events | For the duration of the study (32 weeks)

SECONDARY OUTCOMES:
Number of serious adverse events | For the duration of the study
Number of all adverse events | For the duration of the study
Number of all - daytime and nocturnal - hypoglycaemic events | In the 4 weeks before baseline compared to 4 weeks before interim and final visits
Weight changes compared to baseline | At the end of the study
HbA1c compared to baseline | At the end of the study
Fasting glucose level control compared to baseline as measured by FBG | After 16 and 32 weeks of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Riyadh, Saudi Arabia

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com